CLINICAL TRIAL: NCT01671267
Title: Implementation of Physical Exercise at the Workplace (IRMA06) - Slaughterhouse Workers
Acronym: IRMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre for the Working Environment, Denmark (Other Government)
Responsible Party: Principal Investigator, Lars L. Andersen, Professor, PhD, National Research Centre for the Working Environment, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRMA06
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Musculoskeletal Disorders
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Resistance Training; Ergonomics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Strength training (Experimental): Strength training of the shoulder, arm and hand muscles for 3 x 10 minutes a week.
  Interventions: Behavioral: Strength training
- Ergonomic (Active Comparator): Receives counseling on workstation adjustment and optimal use of the work tools.
  Interventions: Behavioral: Ergonomic

INTERVENTIONS:
Behavioral: Strength training
  Arms: Strength training
Behavioral: Ergonomic
  Arms: Ergonomic

SUMMARY:
The prevalence of pain in the shoulder, arm and hand is high among slaughterhouse workers, allegedly due to the substantial load of these body regions during work. Work disability is a common consequence of these pains. Lowering the physical exposure through ergonomic intervention may be a strategy to reduce the workload. An alternative strategy could be to increase the physical capacity through strength training of the shoulder-, arm- and hand-muscles. This study investigates the effect of two contrasting interventions, i.e. load reduction (ergonomic intervention) versus training of physical capacity (strength training) on pain and work disability in slaughterhouse workers.

The main hypothesis is that strength training intervention for 10 weeks compared with ergonomic intervention results in reduced pain of the shoulder, arm and hand.

ELIGIBILITY:
Inclusion Criteria:

* Slaughterhouse worker
* the pain should have lasted at least 3 months
* pain intensity during the last three months of >= 3 (scale 0-10) in the shoulder, elbow or hand
* the pain should be frequent (at least 3 days per week)

Exclusion Criteria:

* life threatening disease
* pregnancy

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Pain intensity | change from baseline to week 10
  The change in "pain intensity during the last week" (average value of shoulder, elbow and hand) from baseline to 10 week follow-up between the strength training group and ergonomic group. The ergonomic group will be considered the reference group. 2-way analysis of variance (Proc Mixed of SAS) with repeated measures will be used, with time and group as fixed factors and subject as random factor.

SECONDARY OUTCOMES:
DASH | change from baseline to week 10
  Disability of the arm, shoulder and hand questionnaire (DASH). Only the work-module of DASH will be included. Analyzed the same way as the primary outcome.

OTHER OUTCOMES:
PPT | change from baseline to week 10
  Pressure pain threshold of the muscle of the forearm, external rotators of the shoulder, and tibialis anterior of the leg (reference muscle).
WAI | change from baseline to week 10
  Work ability index questionnaire
Total tenderness score | change from baseline to week 10
  change in examiner-verified tenderness of the muscles of the shoulder, arm and hand. Scale of "no", "a little", "moderate" and "severe" tenderness. Summed up to a total tenderness score (Andersen LL 2011, PMID: 21177034)

CONTACTS AND LOCATIONS:
Overall Officials: Lars L Andersen, PhD, Principal Investigator — National Research Centre for the Working Environment, Denmark
Locations (1):
- National Research Centre for the Working Environment, Copenhagen, Denmark

REFERENCES:
- [Derived] Sundstrup E, Jakobsen MD, Brandt M, Jay K, Aagaard P, Andersen LL. Strength Training Improves Fatigue Resistance and Self-Rated Health in Workers with Chronic Pain: A Randomized Controlled Trial. Biomed Res Int. 2016;2016:4137918. doi: 10.1155/2016/4137918. Epub 2016 Oct 17. PMID 27830144
- [Derived] Sundstrup E, Jakobsen MD, Andersen CH, Jay K, Persson R, Aagaard P, Andersen LL. Effect of two contrasting interventions on upper limb chronic pain and disability: a randomized controlled trial. Pain Physician. 2014 Mar-Apr;17(2):145-54. PMID 24658475
- [Derived] Sundstrup E, Jakobsen MD, Andersen CH, Jay K, Persson R, Aagaard P, Andersen LL. Participatory ergonomic intervention versus strength training on chronic pain and work disability in slaughterhouse workers: study protocol for a single-blind, randomized controlled trial. BMC Musculoskelet Disord. 2013 Feb 21;14:67. doi: 10.1186/1471-2474-14-67. PMID 23433448